CLINICAL TRIAL: NCT00046631
Title: Community Characteristics and Physical Activity Among Adolescent Girls
Brief Title: Community Characteristics and Physical Activity Among Adolescent Girls - Ancillary to TAAG
Acronym: TAAG2
Status: Completed | Type: Observational
Sponsor: RAND (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); San Diego State University (Other); University of Minnesota (Other); University of North Carolina, Chapel Hill (Other); University of South Carolina (Other); University of Maryland (Other); University of Arizona (Other); Tulane University (Other)
Responsible Party: Principal Investigator, Deborah Cohen, Sr. Natural Scientist, RAND
Other Study IDs: 1188; R01HL071244 (NIH)
Record Dates: First submitted 2002-09-30; First posted 2002-10-01 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-03

CONDITIONS: Cardiovascular Diseases; Heart Diseases
Keywords: built environment; parks; retail outlets; adolescent girls; physical activity
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adolescent girls: Chosen from 6 schools in 6 cities

SUMMARY:
To investigate the role of community characteristics in physical activity levels of adolescent girls.

DETAILED DESCRIPTION:
BACKGROUND:

The NHLBI-funded multi-centered Trial of Activity for Adolescent Girls (TAAG) is a group (school)-randomized controlled intervention trial to increase physical activity among a cohort of sixth grade girls over 2.5 years.

DESIGN NARRATIVE:

Because environmental factors can influence the likelihood that a person will engage in physical activity, the study investigates the role of community characteristics in physical activity levels. The research forms an ancillary study to the NHLBI-funded multi-centered Trial of Activity for Adolescent Girls (TAAG), a group (school)-randomized controlled intervention trial to increase physical activity among a cohort of sixth grade girls over 2.5 years. The parent TAAG study will be collecting measures of physical activity using both self-report and CSA accelerometers, small monitors worn at the hip that record acceleration and deceleration of movement without the need for any reporting from the participants. Using a radius of 5 miles around each participating TAAG school and around the homes of each study participant, the investigators plan to use geographic information systems (GIS) to gather information documenting proximity of recreational facilities, street design, population density, population mix (ethnic/age distribution), crime, availability of mass transit, neighborhood socioeconomic status (SES), geographic elevations and topography and types of land use. Using hierarchical linear modeling, with girls nested within neighborhoods, while controlling for individual level factors such as race and socioeconomic status, they plan to investigate the relationship of the environment to individual physical activity. In addition, by following girls over time, they plan to investigate whether the effect of the TAAG intervention will be modified by community characteristics. This study will be unique in its scope of exploring the role of community environments in physical activity across six very different urban, suburban, and rural areas: San Diego, CA, Minneapolis, MN, Baltimore, MD, New Orleans, LA, Tucson, AZ and Columbia, SC.

ELIGIBILITY:
No eligibility criteria

Ages: 11 Years to 14 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1556 (Actual)
Dates: Start 2002-08; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Physical activity | 3 years
  We examined the association between built environment features and physical activity

SECONDARY OUTCOMES:
Body Mass Index | 3 years
  We examined the association between built environment features and BMI

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Cohen — RAND
Locations (6):
- United States (6):
  - University of Arizona, Tucson, Arizona
  - San Diego State University, San Diego, California
  - Tulane, New Orleans, Louisiana
  - University of Maryland, Baltimore, Maryland
  - University of Minnesota, Minneapolis, Minnesota
  - University of South Carolina, Columbia, South Carolina

REFERENCES:
- [Result] Scott MM, Cohen DA, Evenson KR, Elder J, Catellier D, Ashwood JS, Overton A. Weekend schoolyard accessibility, physical activity, and obesity: the Trial of Activity in Adolescent Girls (TAAG) study. Prev Med. 2007 May;44(5):398-403. doi: 10.1016/j.ypmed.2006.12.010. Epub 2006 Dec 29. PMID 17292958
- [Result] Cohen DA, Ashwood JS, Scott MM, Overton A, Evenson KR, Staten LK, Porter D, McKenzie TL, Catellier D. Public parks and physical activity among adolescent girls. Pediatrics. 2006 Nov;118(5):e1381-9. doi: 10.1542/peds.2006-1226. PMID 17079539
- [Result] Evenson KR, Scott MM, Cohen DA, Voorhees CC. Girls' perception of neighborhood factors on physical activity, sedentary behavior, and BMI. Obesity (Silver Spring). 2007 Feb;15(2):430-45. doi: 10.1038/oby.2007.502. PMID 17299117
- [Result] Scott MM, Evenson KR, Cohen DA, Cox CE. Comparing perceived and objectively measured access to recreational facilities as predictors of physical activity in adolescent girls. J Urban Health. 2007 May;84(3):346-59. doi: 10.1007/s11524-007-9179-1. PMID 17401691
- [Result] Dowda M, McKenzie TL, Cohen DA, Scott MM, Evenson KR, Bedimo-Rung AL, Voorhees CC, Almeida MJ. Commercial venues as supports for physical activity in adolescent girls. Prev Med. 2007 Aug-Sep;45(2-3):163-8. doi: 10.1016/j.ypmed.2007.06.001. Epub 2007 Jun 7. PMID 17673281